CLINICAL TRIAL: NCT02509676
Title: Effects of Dynamic Stretching Exercise Training on Muscle Tendon Unit
Brief Title: Dynamic Stretching Training and Muscle Tendon Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Funda DEMIRTURK, Asso. Prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-KAEK-097 (Ethics Committee)
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: dynamic stretching training; muscle tendon unit; ultrasound
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dynamic stretching exercise (Experimental): This group will perform dynamic stretching exercise to their left side gastrocnemius muscles for 5 weeks (5 days a week, 3 sets of exercise a day, each set including 5 repetitions of dynamic stretching lasting 45 seconds)
  Interventions: Other: stretching exercise
- control (No Intervention): this group will not perform any stretching exercises for 5 weeks

INTERVENTIONS:
Other: stretching exercise — dynamic stretching exercises with 5 repetitions, each lasting 45 seconds, for 5 days a week and 3 times a day
  Arms: dynamic stretching exercise

SUMMARY:
The purpose of this study is to investigate the effects of a 5-week dynamic stretching exercise training on muscle-tendon unit of gastrocnemius muscle.

DETAILED DESCRIPTION:
Muscle stretching is a common practice applied in warm-up process to enhance performance in sports and to prevent or decrease the risk of sports injury. Muscle stretching is also used for therapeutic purposes in many clinical conditions.

It is generally performed in either static or dynamic manner. The effects of stretching depend on the type, duration and timing of stretching. However, the acute and chronic effects of a stretching can be different in the same muscle.

Recent studies suggest that static stretching has adverse effects on performance, reduces maximal muscle force and is not successful in preventing non-contact injuries, as believed so. Dynamic type is reported to improve flexibility and range of motion better. But there is still debate over which prescription provides the best results in terms of flexibility, power, performance or injury protection. And the answer to the question what happens to the viscoelastic properties of a muscle when it is stretched dynamically for some period of time has not been clearly established.

This study is planned to investigate the effect of a 5-week dynamic stretching exercise training on muscle tendon unit of gastrocnemius muscle. The effects of the training program will be assessed by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Healthy males,
* aged between 18-30 years

Exclusion Criteria:

* Cases with history of recent musculoskeletal injuries or neurological diseases.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
muscle-tendon unit length | at the end of 5 weeks of training
  change in muscle tendon unit property with dynamic exercise training of 5 week will be followed
pennation angle | at the end of 5 weeks of training
  change in pennation angle of the gastrocnemius muscle with dynamic stretching exercise training
muscle thickness | at the end of 5 weeks of training
  change in muscle thickness of the gastrocnemius muscle with dynamic stretching exercise training will be measured by ultrasound

SECONDARY OUTCOMES:
range of ankle dorsiflexion | at the end of 5 weeks of training
  change in range of ankle dorsiflexion with the training program will be assessed with a universal goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Funda DEMIRTURK, PhD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)